CLINICAL TRIAL: NCT06385769
Title: Efficacy of Transcutaneous Tibial Nerve Stimulation in Patients With Neurogenic Overactive Bladder After Stroke: A Randomized Placebo-controlled Clinical Trial.
Brief Title: Transcutaneous Tibial Nerve Stimulation in Patients With Neurogenic Overactive Bladder After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PamukkaleU.ftr-NYıldız-3
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder after stroke; Transcutaneous tibial nerve stimulation; Urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous tibial nerve stimulation (TTNS) (Experimental): In this study, one channel of the stimulation device will provide active stimulation to the patient, while the second channel will not be connected. The patient won't know which channel is active. Both channels will use continuous mode with a pulse frequency of 20 Hz and a pulse width of 200 ms. The intensity for the active channel will be adjusted based on comfort level and observed hallux reaction. Treatment includes 20 sessions of 30 minutes each, administered five times a week for four weeks.
  Interventions: Other: Transcutaneous tibial nerve stimulation (TTNS)
- Sham Transcutaneous tibial nerve stimulation (TTNS) (Sham Comparator): In the placebo group, the same electrotherapy device and settings as the active group will be used. One channel will not be connected to the patient but will display treatment details on the screen. The other channel will be connected but deliver no stimulation. Intensity for the inactive channel is limited to 2-3 mA. Patients will be informed that exceeding this threshold is prevented. Treatment includes 20 sessions of 30 minutes each, administered twice a week for four weeks.
  Interventions: Other: Sham Transcutaneous tibial nerve stimulation (TTNS)

INTERVENTIONS:
Other: Transcutaneous tibial nerve stimulation (TTNS) — The TTNS will be conducted unilaterally, with the patient in a supine position, using a surface electrode dual stimulation channel stimulation device. Two self-adhesive round surface electrodes will be positioned with the negative electrode 2 cm behind the medial malleolus and the positive electrode 10 cm proximal to it. The ground electrode will be placed on the ipsilateral limb. Channel 1 will provide active stimulation, while channel 2 will remain inactive.
  Arms: Transcutaneous tibial nerve stimulation (TTNS)
Other: Sham Transcutaneous tibial nerve stimulation (TTNS) — Sham TTNS group will be stimulated using the same electrotherapy device, with patients positioned identically and electrodes placed in the same positions as in the TTNS group. The current characteristics (pulse frequency 20 Hz and pulse width 200 ms) will also remain consistent across both channels. The second channel of the stimulation device will be designated as the channel connected to the patient but without delivering stimulation.
  Arms: Sham Transcutaneous tibial nerve stimulation (TTNS)

SUMMARY:
The investigators conducted a prospective, randomized, double-blind, placebo-controlled study based on the placebo technique to evaluate the efficacy of TTNS versus placebo in patients with OAB after stroke.

The main questions aimed to be answered are:

What are the effects of Trans Tibial Nerve Stimulation (TTNS) on incontinence-related clinical parameters and quality of life in patients with overactive bladder (OAB) after stroke compared to the placebo group? Participants (n:22) with post-stroke AAM who meet the exclusion and inclusion criteria will be divided into 2 groups using a randomization table. The first group will receive TTNS (n:11) and the second group will receive placebo TTNS (n:11). Measurements will be performed twice in total, before treatment and at the end of treatment (4th week).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 and above with stable ischemic or hemorrhagic stroke.
* Patients with neurogenic detrusor overactivity symptoms accompanied by urinary incontinence complaints and a urinary frequency of 9 or more.
* Patients diagnosed with detrusor overactivity on urodynamic evaluation.
* Patients with hemiplegia lasting between 30 days and 1 year.
* Ability to understand procedures, benefits, and potential side effects.
* Patients scoring 22 or above on the Mini Mental Test.

Exclusion Criteria:

* Patients with post-stroke neurogenic detrusor overactivity receiving or previously received pharmacological treatment.
* Patients using intermittent catheterization or permanent catheterization as a bladder emptying method.
* Patients with a history of urinary incontinence and/or urinary retention before stroke.
* History of past urogynecological surgery.
* Presence of urinary tract infection, bladder tumor, or cardiac pacemaker.
* Significant fluid infusion requirement affecting urination or use of medication affecting bladder function.
* Patients who have received botulinum toxin injection for post-stroke neurogenic detrusor overactivity.
* Patients with postvoid residual volume above 150 mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Decreased frequency of increased voiding | Change from baseline positive response rate at the 4th week after the treatment
  The effectiveness of the treatment is evaluated based on the daily voiding frequency post-treatment compared to the daily voiding frequency pre-treatment. The expected outcome is a reduction in the frequency of increased voiding.

SECONDARY OUTCOMES:
Frequency of voiding | Change from baseline Frequency of voiding, nocturia, number of pads at the 4th week after the treatment
  The frequency of voiding used will be calculated from the patient's 3-day voiding frequency.
The Quality of Life | Change from baseline the Quality of Life at the 4th week after the treatment
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7) will be used to assess specific QoL related to incontinence
Barthel Index for Activities of Daily Living (ADL) | Change from baseline Barthel Index for Activities of Daily Living at the 4th week after the treatment
  The Barthel Index assesses activities of daily living (ADLs), documenting what a patient does daily without determining capabilities. The 10 items to score are: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation, and stair climbing. Scores reflect independence, with lower scores indicating less independence. A score above 60 typically denotes independence.
The Overactive Bladder Symptom Score (OABSS) | Change from baseline The Overactive Bladder Symptom Score at the 4th week after the treatment
  OABSS (Overactive Bladder Symptom Score), four questions assessing daytime frequency (OABSS-1), nocturia frequency (OABSS-2), urgency frequency (OABSS-3), and urgency urinary incontinence (OABSS-4). Severity is rated on a Likert scale from 0-2, 0-3, 0-5, and 0-5, respectively. The total score ranges from 0 to 15, with higher scores indicating more severe symptoms.
Treatment Satisfaction Level | Change from baseline Treatment Satisfaction Level at the 4th week after the treatment
  At the end of the treatment, participants will be asked to evaluate their satisfaction level with the administered treatment using a Likert scale ranging from 1 to 5 (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, 1=very dissatisfied).
Cystometric value | Change from baseline Cystometric value at the 4th week after the treatment
  Cystometric value are useful in defining the voiding characteristics of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin Yıldız, Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas LH, Watkins CL, French B, Sutton C, Forshaw D, Cheater F, Roe B, Leathley MJ, Burton C, McColl E, Booth J; ICONS Project Team; ICONS Patient, Public and Carer Involvement Group. Study protocol: ICONS: identifying continence options after stroke: a randomised trial. Trials. 2011 May 20;12:131. doi: 10.1186/1745-6215-12-131. PMID 21599945
- [Background] Patel M, Coshall C, Rudd AG, Wolfe CD. Natural history and effects on 2-year outcomes of urinary incontinence after stroke. Stroke. 2001 Jan;32(1):122-7. doi: 10.1161/01.str.32.1.122. PMID 11136926
- [Background] Gross T, Schneider MP, Bachmann LM, Blok BF, Groen J, Hoen LA, Castro-Diaz D, Padilla Fernandez B, Del Popolo G, Musco S, Hamid R, Ecclestone H, Karsenty G, Phe V, Pannek J, Kessler TM. Transcutaneous Electrical Nerve Stimulation for Treating Neurogenic Lower Urinary Tract Dysfunction: A Systematic Review. Eur Urol. 2016 Jun;69(6):1102-11. doi: 10.1016/j.eururo.2016.01.010. Epub 2016 Jan 29. PMID 26831506
- [Background] Parittotokkaporn S, Varghese C, O'Grady G, Svirskis D, Subramanian S, O'Carroll SJ. Non-invasive neuromodulation for bowel, bladder and sexual restoration following spinal cord injury: A systematic review. Clin Neurol Neurosurg. 2020 Jul;194:105822. doi: 10.1016/j.clineuro.2020.105822. Epub 2020 Apr 12. PMID 32334284
- [Background] Hagerty JA, Richards I, Kaplan WE. Intravesical electrotherapy for neurogenic bladder dysfunction: a 22-year experience. J Urol. 2007 Oct;178(4 Pt 2):1680-3; discussion 1683. doi: 10.1016/j.juro.2007.03.188. Epub 2007 Aug 17. PMID 17707024
- [Background] Nardone R, Versace V, Sebastianelli L, Brigo F, Golaszewski S, Christova M, Saltuari L, Trinka E. Transcranial magnetic stimulation and bladder function: A systematic review. Clin Neurophysiol. 2019 Nov;130(11):2032-2037. doi: 10.1016/j.clinph.2019.08.020. Epub 2019 Sep 3. PMID 31541980
- [Background] Araujo TG, Schmidt AP, Sanches PRS, Silva Junior DP, Rieder CRM, Ramos JGL. Transcutaneous tibial nerve home stimulation for overactive bladder in women with Parkinson's disease: A randomized clinical trial. Neurourol Urodyn. 2021 Jan;40(1):538-548. doi: 10.1002/nau.24595. Epub 2020 Dec 16. PMID 33326648
- [Background] Perissinotto MC, D'Ancona CA, Lucio A, Campos RM, Abreu A. Transcutaneous tibial nerve stimulation in the treatment of lower urinary tract symptoms and its impact on health-related quality of life in patients with Parkinson disease: a randomized controlled trial. J Wound Ostomy Continence Nurs. 2015 Jan-Feb;42(1):94-9. doi: 10.1097/WON.0000000000000078. PMID 25549314
- [Background] Gaspard L, Tombal B, Opsomer RJ, Castille Y, Van Pesch V, Detrembleur C. [Physiotherapy and neurogenic lower urinary tract dysfunction in multiple sclerosis patients: a randomized controlled trial]. Prog Urol. 2014 Sep;24(11):697-707. doi: 10.1016/j.purol.2014.05.003. Epub 2014 Jun 19. French. PMID 25214451
- [Background] Zonic-Imamovic M, Imamovic S, Cickusic A, Delalic A, Hodzic R, Imamovic M. Effects of Treating an Overactive Urinary Bladder in Patients with Multiple Sclerosis. Acta Med Acad. 2019 Dec;48(3):271-277. doi: 10.5644/ama2006-124.267. PMID 32124625
- [Background] Eftekhar T, Teimoory N, Miri E, Nikfallah A, Naeimi M, Ghajarzadeh M. Posterior tibial nerve stimulation for treating neurologic bladder in women: a randomized clinical trial. Acta Med Iran. 2014;52(11):816-21. PMID 25415813
- [Background] Monteiro ES, de Carvalho LB, Fukujima MM, Lora MI, do Prado GF. Electrical stimulation of the posterior tibialis nerve improves symptoms of poststroke neurogenic overactive bladder in men: a randomized controlled trial. Urology. 2014 Sep;84(3):509-14. doi: 10.1016/j.urology.2014.05.031. PMID 25168524
- [Background] Liu Y, Xu G, Luo M, Teng HF. Effects of Transcutaneous Electrical Nerve Stimulation at Two Frequencies on Urinary Incontinence in Poststroke Patients: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2016 Mar;95(3):183-93. doi: 10.1097/PHM.0000000000000360. PMID 26259053
- [Background] Erden E, Ersoz M, Erden E, Tiftik T. Urodynamic findings and therapeutic approaches for neurogenic lower urinary tract dysfunction in patients with thoracic spinal cord injury. Ir J Med Sci. 2023 Oct;192(5):2513-2520. doi: 10.1007/s11845-022-03239-9. Epub 2022 Dec 1. PMID 36454536
- [Background] Booth J, Hagen S, McClurg D, Norton C, MacInnes C, Collins B, Donaldson C, Tolson D. A feasibility study of transcutaneous posterior tibial nerve stimulation for bladder and bowel dysfunction in elderly adults in residential care. J Am Med Dir Assoc. 2013 Apr;14(4):270-4. doi: 10.1016/j.jamda.2012.10.021. Epub 2012 Nov 30. PMID 23206722
- [Background] Schreiner L, dos Santos TG, Knorst MR, da Silva Filho IG. Randomized trial of transcutaneous tibial nerve stimulation to treat urge urinary incontinence in older women. Int Urogynecol J. 2010 Sep;21(9):1065-70. doi: 10.1007/s00192-010-1165-6. Epub 2010 May 11. PMID 20458465
- [Background] Ozerdogan N, Beji NK, Yalcin O. Urinary incontinence: its prevalence, risk factors and effects on the quality of life of women living in a region of Turkey. Gynecol Obstet Invest. 2004;58(3):145-50. doi: 10.1159/000079422. Epub 2004 Jun 29. PMID 15237249
- [Background] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723
- [Background] Culha MG, Degirmentepe RB, Ozbir S, Cakir SS, Homma Y. Turkish validation of the overactive bladder symptom score (OABSS) and evaluation of mirabegron treatment response. Int Urogynecol J. 2019 Dec;30(12):2121-2126. doi: 10.1007/s00192-019-04054-0. Epub 2019 Jul 22. PMID 31332467
- [Background] Kim SJ, Choi HW, Cho HJ, Hwang TK, Kim JC. The influence of preoperative bladder outlet obstruction on continence and satisfaction in patients with stress urinary incontinence after midurethral sling. Int Neurourol J. 2010 Dec;14(4):267-71. doi: 10.5213/inj.2010.14.4.267. Epub 2010 Dec 31. PMID 21253340